CLINICAL TRIAL: NCT00744237
Title: Glycemic Effects of Nebivolol Compared With Metoprolol Extended Release and Compared With Hydrochlorothiazide In Hypertensive Patients With Type 2 Diabetes Mellitus: A Pilot Study
Brief Title: Study of the Glycemic Effects of Nebivolol Compared With Metoprolol and HCTZ in Diabetic Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: John Whalen, MD, Executive Director, Clinical Development, Cardiovascular, Forest Research Institute, a Subsidiary of Forest Laboratories Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-19
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus
Keywords: nebivolol; Bystolic ™; Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Nebivolol; Metoprolol; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): * Nebivolol 5 mg (overencapsulated 5-mg marketed tablet), oral administration
  * Nebivolol 10 mg (overencapsulated 10-mg marketed tablet), oral administration
  * Nebivolol 20 mg (overencapsulated 20-mg marketed tablet) oral administration
  * Nebivolol 40 mg (two overencapsulated 20-mg tablets) oral administration
  * Open-label amlodipine may be given
  Interventions: Drug: Nebivolol
- 2 (Active Comparator): * Metoprolol ER 50 mg (overencapsulated 50-mg tablet) oral administration
  * Metoprolol ER 100 mg (two overencapsulated 50-mg tablets) oral administration
  * Metoprolol ER 200 mg (overencapsulated 200-mg tablet) oral administration
  * Metoprolol ER 400 mg (two overencapsulated 200-mg tablets) oral administration
  * Open-label amlodipine may be given
  Interventions: Drug: Metoprolol ER
- 3 (Active Comparator): * HCTZ 12.5 mg (overencapsulated 12.5 capsule), oral administration
  * HCTZ 25 mg (two capsules, overencapsulated 12.5-mg capsules), oral administration
  * Open-label amlodipine may be given
  Interventions: Drug: HCTZ

INTERVENTIONS:
Drug: Nebivolol — * Nebivolol 5 mg (overencapsulated 5-mg marketed tablet), oral administration
  * Nebivolol 10 mg (overencapsulated 10-mg marketed tablet), oral administration
  * Nebivolol 20 mg (overencapsulated 20-mg marketed tablet) oral administration
  * Nebivolol 40 mg (two overencapsulated 20-mg tablets) oral administration
  Other Names: Bystolic (TM)
  Arms: 1
Drug: Metoprolol ER — * Metoprolol ER 50 mg (overencapsulated 50-mg tablet) oral administration
  * Metoprolol ER 100 mg (two overencapsulated 50-mg tablets) oral administration
  * Metoprolol ER 200 mg (overencapsulated 200-mg tablet) oral administration
  * Metoprolol ER 400 mg (two overencapsulated 200-mg tablets) oral administration
  Arms: 2
Drug: HCTZ — * HCTZ 12.5 mg (overencapsulated 12.5 capsule), oral administration
  * HCTZ 25 mg (two capsules, overencapsulated 12.5-mg capsules), oral administration
  Other Names: Hydrochlorothorazide
  Arms: 3

SUMMARY:
This study will evaluate the effects of nebivolol on glycemic control compared with metoprolol and HCTZ in patients with hypertension and type 2 diabetes mellitus

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female, 18-85 years of age
* Blood pressure in the range of 130 to 179/80 to 109 mmHg
* Currently using either an ACE inhibitor or an ARB alone or (an ACE inhibitor or an ARB and up to two other drugs for treatment of high blood pressure). (Patients may be on both an ACE inhibitor and ARB, but would need to be taken off one.)
* Stable medication regimen for high blood pressure for at least one month prior to screening
* Stable type 2 diabetes mellitus for at least 3 months prior to screening that is controlled by any or all of the following: diet and antidiabetic medications that may include fixed-dose insulin
* HgbA1c 6.5 to 8.5% (This is measured at the screening visit)

EXCLUSION CRITERIA:

* Use of any beta blocker within one month prior to screening
* Use of clonidine within 3 months prior to screening
* Diagnosis of hyperthyroidism as evidenced by abnormal lab markers
* Any disorder requiring the intermittent or chronic use of systemic corticosteroids
* Diagnosis of hyperthyroidism as determined by lab markers done at screening
* Active liver disease as determined by lab markers
* Kidney impairment; estimated GFR < 60 mL/min/1.73 m2
* History of heart attack, clinically significant arrhythmia, unstable angina, coronary angioplasty/bypass surgery, stroke, or TIA in 3 months prior to screening
* Chronic heart failure
* Drug or alcohol abuse within 2 years prior to screening
* History of sensitivity to any beta blocker, HCTZ, sulfa drug, or calcium channel blocker
* Participation in another research study within 30 days prior to screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Shea, MS, Study Director — Forest Research Institute, a Subsidiary of Forest Laboratories, Inc.
Locations (65):
- United States (62):
  - Forest Investigative Site 15, Athens, Alabama
  - Forest Investigative Site 16, Huntsville, Alabama
  - Forest Investigative Site 35, Bell Gardens, California
  - Forest Investigative Site, Buena Park, California
  - Forest Investigative Site 54, Chino, California
  - Forest Investigative Site 40, Fremont, California
  - Forest Investigative Site, Palm Springs, California
  - Forest Investigative Site, Pomona, California
  - Forest Investigative Site 55, Sacramento, California
  - Forest Investigative Site 11, San Diego, California
  - Forest Investigative Site, Santa Monica, California
  - Forest Investigative Site, Spring Valley, California
  - Forest Investigative Site 49, Tustin, California
  - Forest Investigative Site 47, Walnut Creek, California
  - Forest Investigative Site 61, Golden, Colorado
  - Forest Investigative Site, Wheat Ridge, Colorado
  - Forest Investigative Site 3, Daytona Beach, Florida
  - Forest Investigative Site 33, DeLand, Florida
  - Forest Investigative Site 36, Hollywood, Florida
  - Forest Investigative Site 62, Miami, Florida
  - Forest Investigative Site 080, Miami, Florida
  - Forest Investigative Site 59, Miami, Florida
  - Forest Investigative Site 32, Pembroke Pines, Florida
  - Forest Investigative Site 081, Pembroke Pines, Florida
  - Forest Investigative Site 2, Tamarac, Florida
  - Forest Investigative Site, Tampa, Florida
  - Forest Investigative Site 19, West Palm Beach, Florida
  - Forest Investigative Site 44, Atlanta, Georgia
  - Forest Investigative Site 5, Augusta, Georgia
  - Forest Investigative Site 56, Honolulu, Hawaii
  - Forest Investigative Site 57, Meridian, Idaho
  - Forest Investigative Site 39, Chicago, Illinois
  - Forest Investigative Site 37, Wichita, Kansas
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site 20, Baltimore, Maryland
  - Forest Investigative Site 50, Oxon Hill, Maryland
  - Forest Investigative Site 21, Saint Clair Shores, Michigan
  - Forest Investigative Site, Kansas City, Missouri
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, New Hyde Park, New York
  - Forest Investigative Site, New York, New York
  - Forest Investigative Site 7, Charlotte, North Carolina
  - Forest Investigative Site 45, Charlotte, North Carolina
  - Forest Investigative Site 24, Morehead City, North Carolina
  - Forest Investigative Site 26, Salisbury, North Carolina
  - Forest Investigative Site 18, Wilmington, North Carolina
  - Forest Investigative Site 51, Centerville, Ohio
  - Forest Investigative Site 48, Cincinnati, Ohio
  - Forest Investigative Site 12, Wadsworth, Ohio
  - Forest Investigative Site 17, Charleston, South Carolina
  - Forest Investigative Site 46, Columbia, South Carolina
  - Forest Investigative Site, North Charleston, South Carolina
  - Forest Investigative Site, Simpsonville, South Carolina
  - Forest Investigative Site 4, Sioux Falls, South Dakota
  - Forest Investigative Site 10, New Tazewell, Tennessee
  - Forest Investigative Site 52, Corpus Christi, Texas
  - Forest Investigative Site 28, Dallas, Texas
  - Forest Investigative Site 38, Hurst, Texas
  - Forest Investigative Site 34, Salt Lake City, Utah
  - Forest Investigative Site, St. George, Utah
  - Forest Investigative Site, Norfolk, Virginia
  - Forest Investigative Site 31, Virginia Beach, Virginia
- Puerto Rico (3):
  - Forest Investigative Site 41, Ponce
  - Forest Investigative Site 60, Salinas
  - Forest Investigative Site 29, Santurce

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured from September 2008 through December 2009 at 69 US sites
Pre-assignment Details: Placebo washout phase was required for patients currently on any anti-hypertensives at screening exclusive of background ACE inhibitor or ARB before assignment to HCTZ or Metoprolol ER or Nebivolol arms.
Groups:
- Nebivolol: * Nebivolol 5 mg (overencapsulated 5-mg marketed tablet), oral administration
  * Nebivolol 10 mg (overencapsulated 10-mg marketed tablet), oral administration
  * Nebivolol 20 mg (overencapsulated 20-mg marketed tablet) oral administration
  * Nebivolol 40 mg (two overencapsulated 20-mg tablets) oral administration
  * Open-label amlodipine may be given
- Metoprolol ER: * Metoprolol ER 50 mg (overencapsulated 50-mg tablet) oral administration
  * Metoprolol ER 100 mg (two overencapsulated 50-mg tablets) oral administration
  * Metoprolol ER 200 mg (overencapsulated 200-mg tablet) oral administration
  * Metoprolol ER 400 mg (two overencapsulated 200-mg tablets) oral administration
  * Open-label amlodipine may be given
- Hydrochlorothiazide (HCTZ): * HCTZ 12.5 mg (overencapsulated 12.5 capsule), oral administration
  * HCTZ 25 mg (two capsules, overencapsulated 12.5-mg capsules), oral administration
  * Open-label amlodipine may be given
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol ER | Hydrochlorothiazide (HCTZ)
Started | 83 | 73 | 74
Completed | 56 | 46 | 59
Not Completed | 27 | 27 | 15
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Protocol Violation | 3 | 4 | 3
Not completed — Inclusion/Exclusion criteria not met | 1 | 0 | 0
Not completed — Dosing Error | 1 | 0 | 1
Not completed — Study Drug Error | 1 | 0 | 0
Not completed — Prohibited Concomitant Medication | 0 | 0 | 1
Not completed — Poor Compliance | 0 | 2 | 0
Not completed — Administrative. Site Closed | 1 | 1 | 1
Not completed — Adverse Event | 9 | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol ER | Hydrochlorothiazide (HCTZ) | Total
Number analyzed (Participants) | 83 | 73 | 74 | 230
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.3) | 59.2 (8.3) | 59.5 (9.0) | 58.9 (8.9)
Age, Customized [Number; unit: participants]
  Patients 18 to 64 years of age | 61 | 51 | 53 | 165
  Patients greater than or equal to 65 years of age. | 22 | 22 | 21 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 29 | 89
  Male | 53 | 43 | 45 | 141
Region of Enrollment [Number; unit: participants]
  United States | 78 | 69 | 72 | 219
  Puerto Rico | 5 | 4 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Glycosylated Hemoglobin (HbA1c) at Week 26
Description: Change from baseline in glycosylated hemoglobin (HbA1c) over 26 weeks, Last Observation Carried Forward.
Time Frame: visit 5(week 0) and visit 14(week 26)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nebivolol | Metoprolol ER | Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 77 | 69 | 68
Percentage | 0.12 (0.78) | 0.00 (0.65) | 0.40 (0.96)

2. Secondary Outcome: Change From Baseline in Insulin Resistance Based on Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Change from Baseline in Insulin Resistance based on homeostasis model assessment of insulin resistance (HOMA-IR) at week 26, Last Observation Carried Forward (LOCF). The HOMA-IR is the the product of the blood Glucose and Insulin levels, divided by a constant. HOMA-IR is expressed as the following: HOMA-IR = fasting serum insulin (μU/ml) × fasting plasma glucose (mmol/l) / 22.5
Time Frame: [visit 5(week 0) and visit 14(week 26)]
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Nebivolol | Metoprolol ER | Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 77 | 69 | 68
Unit on a scale | 0.011 (9.828) | 1.156 (9.628) | -0.662 (10.178)

ADVERSE EVENTS:
Time Frame: Adverse Events were reported over a 12-month period, from September 2008 to August 2010.
Arm/Group | Nebivolol | Metoprolol ER | Hydrochlorothiazide (HCTZ)
Serious Adverse Events (participants affected / at risk) | 2/83 | 3/73 | 2/74
Other Adverse Events (participants affected / at risk) | 19/83 | 17/73 | 17/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=83) | Metoprolol ER (N=73) | Hydrochlorothiazide (HCTZ) (N=74)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0
Deep vain thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Incision site cellulitis (Infections and infestations) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=83) | Metoprolol ER (N=73) | Hydrochlorothiazide (HCTZ) (N=74)
Bradycardia (Cardiac disorders) | 6 | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1
Dizziness (Nervous system disorders) | 5 | 3 | 3
Fatigue (General disorders) | 3 | 1 | 5
Headache (Nervous system disorders) | 5 | 7 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 5
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3
Oedema peripheral (General disorders) | 8 | 7 | 6
Upper Resiratory tract infection (Infections and infestations) | 2 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute.